CLINICAL TRIAL: NCT03412552
Title: Risk Analysis of Intensive Care Management on Maternal and Fetal Outcome of Severe Preeclampsia and Eclampsia
Brief Title: Risk Analysis of Intensive Care Mangement on Maternal and Fetal Outcome of Severe Preeclampsia and Eclampsia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 22
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Toxemia | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- severe preeclampsia without HELLP syndrome: severe preeclampsia if they met one or more of the following criteria of The American College of Obstetricians and Gynecologists (10): systolic blood pressure >160 mm/ Hg or diastolic blood pressure >110 mm/Hg, headache, epigastric or right-upper-quadrant pain, visual disturbances,pulmonary edema, and proteinuria (urinary protein level >5 g/24 h).Women with severe preeclampsia selected for analysis also met all of the following laboratory criteria: platelet count ≥150,000/ mm3, serum lactate dehydrogenase <600 IU /dL, serum total bilirubin <1.2 mg/dL and serum aspartate aminotransferase <70IU/L
  Interventions: Drug: MgSO4
- eclampsia without HELLP syndrome: Eclampsia was defined as tonic-clonic seizures occurring in patient diagnosed by preeclampsia patient. Any causes for convulsion other than eclampsia were excluded
  Interventions: Drug: MgSO4
- eclampsia with HELLP syndrome: Eclampsia was defined as tonic-clonic seizures occurring in patient diagnosed by preeclampsia patient. Any causes for convulsion other than eclampsia were excluded.HELLP syndrome was defined by the clinical presentation of PET in association with thrombocytopenia (<150.000 cells/ul), hemolysis and elevated liver enzmes (elevated transaminases and lactic dyhydrogenases activities)
  Interventions: Drug: MgSO4
- HELLP syndrome without eclampsia: HELLP syndrome was defined by the clinical presentation of PET in association with thrombocytopenia (<150.000 cells/ul), hemolysis and elevated liver enzmes (elevated transaminases and lactic dyhydrogenases activities)
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: MgSO4 — Loading dose of magensium sulphate (4-6g I.V), given over 20 minutes in 100 ml of dextrose, Maintenance dose (4-6g) magensium sulphate in 500 cc dextrose given over 8 hours using continuous IV drip
  Other Names: magnesium Sulfate

SUMMARY:
Laboratory monitoring of patients included serial measurement of complete blood cell count, liver function tests, coagulation profile, and renal function tests.

ICU management during conduction of the research study included the following:

Control of convulsions using magensium sulphate. Control of blood pressure Diastolic blood pressure above 110 mmHg, nifedipine was administered.A plasma volume expansion with saline was used in all women to maintain sufficient intravascular volume. Delivery was performed immediately after hemodynamic stabilization and clinical control of general condition .

DETAILED DESCRIPTION:
Laboratory monitoring of patients included serial measurement of complete blood cell count, liver function tests, coagulation profile, and renal function tests.

ICU management included the following:

Control of convulsions by Loading dose of magensium sulphate (4-6g I.V), given over 20 minutes in 100 ml of dextrose then Maintenance dose (4-6g) magensium sulphate in 500 cc dextrose given over 8 hours using continuous IV drip.Control of blood pressure if Diastolic blood pressure above 110 mmHg, nifedipine was administered. Delivery was performed immediately after hemodynamic stabilization and clinical control of general condition .Termination of gestation decision was based on the the presence of maternal complications, fetal distress.After delivery the patient is retrurned to ICU under clinical and careful observation of the following:Heart rate, blood pressure,every 15 min,Temperature and respiratory rate ,evey 4 hours. Duration of admission in the ICU was assessed

ELIGIBILITY:
Inclusion Criteria:

* women with severe preeclampsia or eclampsia or HELLP syndrome admitted to ICU

Exclusion Criteria:

Non eclamptic causes of fits, including hysterical causes and epilepsy

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients were diagnosed as severe preeclampsia if met one or more of the American College of Obstetricians and Gynecologists Eclampsia was defined as tonic-clonic seizures occurring in patient diagnosed by preeclampsia patient. .HELLP syndrome was defined by the clinical presentation of PET in association with thrombocytopenia (<150.000 cells/ul), hemolysis and elevated liver enzmes (elevated transaminases and lactic dyhydrogenases activities).
Sampling Method: Non-Probability Sample
Enrollment: 1238 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
control of blood pressure | 24 hours after delivery
  keeping blood pressure at or below 140/90

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided